CLINICAL TRIAL: NCT01673867
Title: An Open-Label Randomized Phase III Trial of BMS-936558 (Nivolumab) Versus Docetaxel in Previously Treated Metastatic Non-squamous Non-small Cell Lung Cancer (NSCLC)
Brief Title: Study of BMS-936558 (Nivolumab) Compared to Docetaxel in Previously Treated Metastatic Non-squamous NSCLC
Acronym: CheckMate057
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-057; 2012-002472-14 (EudraCT Number)
Expanded Access: NCT03126643 (Approved for marketing)
Record Dates: First submitted 2012-08-24; First posted 2012-08-28 (Estimated); Results first posted 2016-02-26 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Non-Squamous Cell Non-small Cell Lung Cancer
MeSH Terms: interventions — Nivolumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Nivolumab (Experimental): Nivolumab 3 mg/kg solution intravenously (IV) every 2 weeks until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends. Eligible patients may receive nivolumab at 480mg every 4 weeks until documented disease progression, discontinuation, withdrawal of consent or the study ends.
  Interventions: Biological: Nivolumab
- Arm B: Docetaxel (Active Comparator): Docetaxel 75 mg/m^2 concentrate for solution for intravenous infusion every 3 weeks until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends. Eligible patients may receive nivolumab at 480mg every 4 weeks until documented disease progression, discontinuation, withdrawal of consent or the study ends.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Biological: Nivolumab
  Other Names: BMS-936558 (Anti-PD1)
  Arms: Arm A: Nivolumab
Drug: Docetaxel
  Other Names: Taxotere®
  Arms: Arm B: Docetaxel

SUMMARY:
The purpose of the study is to compare the overall survival of BMS-936558 (Nivolumab) as compared with Docetaxel in subjects with non-squamous cell non-small cell lung cancer (NSCLC) after failure of prior platinum-based chemotherapy

DETAILED DESCRIPTION:
CheckMate 057: CHECKpoint pathway and nivoluMAb clinical Trial Evaluation 057

ELIGIBILITY:
Inclusion Criteria:

* Men & women ≥18 years of age
* Subjects with histologically or cytologically-documented non-squamous cell NSCLC who present with Stage IIIB/IV disease or recurrent or progressive disease following multimodal therapy (radiation therapy, surgical resection, or definitive chemoradiation therapy for locally advanced disease) and who will receive study therapy as second or third line of treatment for advanced disease
* Disease recurrence or progression during/after one prior platinum doublet-based chemotherapy regimen for advanced or metastatic disease
* Measurable disease by Computed tomography (CT)/Magnetic resonance imaging (MRI) per RECIST 1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1
* A formalin fixed, paraffin-embedded (FFPE) tumor tissue block or unstained slides of tumor sample (archival or recent) must be available for biomarker evaluation. Specimens must be received by the central lab prior to randomization. Biopsy should be excisional, incisional or core needle. Fine needle aspiration is insufficient

Exclusion Criteria:

* Subjects with untreated central nervous system (CNS) metastases are excluded. Subjects are eligible if CNS metastases are asymptomatic or treated and subjects are neurologically returned to baseline for at least 2 weeks prior to enrollment. In addition, subjects must be either off corticosteroids, or on a stable or decreasing dose of ≤10mg daily prednisone (or equivalent)
* Subjects with carcinomatous meningitis
* Subjects with active or recent history of known or suspected autoimmune disease. Subjects with Type 1 diabetes mellitus, hypothyroidism only requiring hormone replacement, or skin disorders (vitiligo, psoriasis, or alopecia) not requiring systemic treatment are permitted to enroll
* Subjects with a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days of randomization
* Prior therapy with anti-programmed death-1 (anti-PD-1), anti-programmed cell death ligand 1 (anti-PD-L1), anti-programmed cell death ligand 2 (anti-PD-L2), anti-cluster of differentiation 137 (anti-CD137), or anti-Cytotoxic T lymphocyte-associated antigen 4 (anti-CTLA-4) antibody (including Ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Prior treatment with Docetaxel
* Treatment with any investigational agent within 14 days of first administration of study treatment

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 582 (Actual)
Dates: Start 2012-11-02 (Actual); Primary Completion 2015-02-05 (Actual); Study Completion 2021-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (117):
- United States (30):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Local Institution - 0009, Duarte, California
  - Local Institution - 0042, San Diego, California
  - San Francisco Oncology Associates, San Francisco, California
  - Yale University, New Haven, Connecticut
  - Local Institution - 0034, Tampa, Florida
  - Northwest Georgia Oncology Center, P.C., Marietta, Georgia
  - Local Institution - 0030, Chicago, Illinois
  - The Johns Hopkins University, Baltimore, Maryland
  - Local Institution - 0031, Boston, Massachusetts
  - Local Institution - 0040, Boston, Massachusetts
  - Local Institution - 0138, Boston, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Local Institution - 0008, Mineola, New York
  - Local Institution - 0020, New York, New York
  - Local Institution - 0027, Durham, North Carolina
  - Local Institution - 0026, Cincinnati, Ohio
  - St. Mary Medical Center, Langhorne, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Local Institution - 0035, Sayre, Pennsylvania
  - Local Institution - 0025, Columbia, South Carolina
  - Local Institution - 0024, Chattanooga, Tennessee
  - Local Institution - 0028, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Local Institution - 0033, Dallas, Texas
  - Local Institution - 0032, Houston, Texas
  - Local Institution - 0041, Kennewick, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Local Institution - 0007, Seattle, Washington
  - Local Institution - 0019, Morgantown, West Virginia
- Argentina (5):
  - Local Institution - 0010, Capital Federal, Buenos Aires
  - Local Institution - 0057, Capital Federal, Buenos Aires
  - Local Institution - 0124, Ciudad de Buenos Aires, Buenos Aires
  - Local Institution - 0011, Buenos Aires
  - Local Institution - 0125, La Rioja
- Australia (6):
  - Local Institution, Tweed Heads, New South Wales
  - Local Institution, Woolloongabba, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, Kurralta Park, South Australia
  - Local Institution, Frankston, Victoria
  - Local Institution, Melbourne, Victoria
- Austria (4):
  - Local Institution, Linz
  - Local Institution, Salzburg
  - Local Institution, Vienna
  - Local Institution, Wels
- Brazil (6):
  - Local Institution - 0056, Fortaleza, Ceará
  - Local Institution - 0054, Salvador, Estado de Bahia
  - Local Institution - 0053, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0055, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0052, Barretos, São Paulo
  - Local Institution - 0051, Rio de Janeiro
- Canada (3):
  - Local Institution - 0133, Edmonton, Alberta
  - Local Institution, London, Ontario
  - Local Institution - 0110, Rimouski, Quebec
- Chile (4):
  - Local Institution - 0012, Viña del Mar, Región de Valparaíso
  - Local Institution - 0058, Santiago, Santiago Metropolitan
  - Local Institution - 0077, Santiago, Santiago Metropolitan
  - Local Institution - 0134, Santiago, Santiago Metropolitan
- Local Institution - 0018, Prague, Czechia
- France (8):
  - Local Institution, Créteil
  - Local Institution, Dijon
  - Local Institution - 0119, La Roche-sur-Yon
  - Local Institution - 0113, Lyon
  - Local Institution - 0112, Marseille
  - Local Institution, Poitiers
  - Local Institution - 0114, Rennes
  - Local Institution, Toulouse
- Germany (8):
  - Local Institution, Bad Berka
  - Local Institution - 0090, Cologne
  - Local Institution, Großhansdorf
  - Local Institution, Heidelberg
  - Local Institution, Mainz
  - Local Institution, Recklinghausen
  - Local Institution, Stuttgart
  - Local Institution, Ulm
- Hong Kong (2):
  - Local Institution - 0043, Hong Kong
  - Local Institution, Hong Kong
- Local Institution - 0074, Budapest, Hungary
- Italy (9):
  - Local Institution - 0122, Bergamo
  - Local Institution - 0086, Bologna
  - Local Institution - 0087, Meldola (fc)
  - Local Institution - 0085, Milan
  - Local Institution - 0084, Padua
  - Local Institution - 0121, Parma
  - Local Institution - 0083, Perugia
  - Local Institution - 0088, Ravenna
  - Local Institution - 0082, Siena
- Mexico (4):
  - Local Institution - 0107, Mexico City, Mexico City
  - Local Institution - 0108, Mexico City, Mexico City
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Hermosillo, Sonora
- Local Institution - 0141, Oslo, Norway
- Peru (4):
  - Local Institution - 0131, Miraflores, Lima region
  - Local Institution - 0050, Arequipa
  - Local Institution - 0048, Lima
  - Local Institution - 0049, Lima
- Poland (5):
  - Local Institution - 0073, Krakow, Lesser Poland Voivodeship
  - Local Institution - 0068, Gdansk
  - Local Institution - 0072, Olsztyn
  - Local Institution - 0067, Szczecin
  - Local Institution - 0070, Warsaw
- Romania (5):
  - Local Institution - 0099, Bucharest
  - Local Institution - 0123, Cluj-Napoca
  - Local Institution - 0063, Craiova
  - Local Institution - 0061, Iași
  - Local Institution - 0062, Timișoara
- Russia (4):
  - Local Institution - 0078, Moscow
  - Local Institution - 0079, Moscow
  - Local Institution - 0120, Moscow
  - Local Institution - 0080, Saint Petersburg
- Local Institution, Singapore, Singapore
- Spain (4):
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution - 0001, Seville
  - Local Institution, Vizcaya
- Switzerland (2):
  - Local Institution, Basel
  - Local Institution, Chur

REFERENCES:
- [Derived] Barrera C, Corredor G, Viswanathan VS, Ding R, Toro P, Fu P, Buzzy C, Lu C, Velu P, Zens P, Berezowska S, Belete M, Balli D, Chang H, Baxi V, Syrigos K, Rimm DL, Velcheti V, Schalper K, Romero E, Madabhushi A. Deep computational image analysis of immune cell niches reveals treatment-specific outcome associations in lung cancer. NPJ Precis Oncol. 2023 Jun 1;7(1):52. doi: 10.1038/s41698-023-00403-x. PMID 37264091
- [Derived] Hu S, Tang Z, Harrison JP, Hertel N, Penrod JR, May JR, Juarez-Garcia A, Holdgate O. Economic Evaluation of Nivolumab Versus Docetaxel for the Treatment of Advanced Squamous and Non-squamous Non-small Cell Lung Cancer After Prior Chemotherapy in China. Pharmacoecon Open. 2023 Mar;7(2):273-284. doi: 10.1007/s41669-022-00383-x. Epub 2023 Mar 10. PMID 36897427
- [Derived] Borghaei H, Gettinger S, Vokes EE, Chow LQM, Burgio MA, de Castro Carpeno J, Pluzanski A, Arrieta O, Frontera OA, Chiari R, Butts C, Wojcik-Tomaszewska J, Coudert B, Garassino MC, Ready N, Felip E, Garcia MA, Waterhouse D, Domine M, Barlesi F, Antonia S, Wohlleber M, Gerber DE, Czyzewicz G, Spigel DR, Crino L, Eberhardt WEE, Li A, Marimuthu S, Brahmer J. Five-Year Outcomes From the Randomized, Phase III Trials CheckMate 017 and 057: Nivolumab Versus Docetaxel in Previously Treated Non-Small-Cell Lung Cancer. J Clin Oncol. 2021 Mar 1;39(7):723-733. doi: 10.1200/JCO.20.01605. Epub 2021 Jan 15. PMID 33449799
- [Derived] Long GV, Tykodi SS, Schneider JG, Garbe C, Gravis G, Rashford M, Agrawal S, Grigoryeva E, Bello A, Roy A, Rollin L, Zhao X. Assessment of nivolumab exposure and clinical safety of 480 mg every 4 weeks flat-dosing schedule in patients with cancer. Ann Oncol. 2018 Nov 1;29(11):2208-2213. doi: 10.1093/annonc/mdy408. PMID 30215677
- [Derived] Reck M, Brahmer J, Bennett B, Taylor F, Penrod JR, DeRosa M, Dastani H, Spigel DR, Gralla RJ. Evaluation of health-related quality of life and symptoms in patients with advanced non-squamous non-small cell lung cancer treated with nivolumab or docetaxel in CheckMate 057. Eur J Cancer. 2018 Oct;102:23-30. doi: 10.1016/j.ejca.2018.05.005. Epub 2018 Aug 10. PMID 30103096
- [Derived] Vokes EE, Ready N, Felip E, Horn L, Burgio MA, Antonia SJ, Aren Frontera O, Gettinger S, Holgado E, Spigel D, Waterhouse D, Domine M, Garassino M, Chow LQM, Blumenschein G Jr, Barlesi F, Coudert B, Gainor J, Arrieta O, Brahmer J, Butts C, Steins M, Geese WJ, Li A, Healey D, Crino L. Nivolumab versus docetaxel in previously treated advanced non-small-cell lung cancer (CheckMate 017 and CheckMate 057): 3-year update and outcomes in patients with liver metastases. Ann Oncol. 2018 Apr 1;29(4):959-965. doi: 10.1093/annonc/mdy041. PMID 29408986
- [Derived] Horn L, Spigel DR, Vokes EE, Holgado E, Ready N, Steins M, Poddubskaya E, Borghaei H, Felip E, Paz-Ares L, Pluzanski A, Reckamp KL, Burgio MA, Kohlhaeufl M, Waterhouse D, Barlesi F, Antonia S, Arrieta O, Fayette J, Crino L, Rizvi N, Reck M, Hellmann MD, Geese WJ, Li A, Blackwood-Chirchir A, Healey D, Brahmer J, Eberhardt WEE. Nivolumab Versus Docetaxel in Previously Treated Patients With Advanced Non-Small-Cell Lung Cancer: Two-Year Outcomes From Two Randomized, Open-Label, Phase III Trials (CheckMate 017 and CheckMate 057). J Clin Oncol. 2017 Dec 10;35(35):3924-3933. doi: 10.1200/JCO.2017.74.3062. Epub 2017 Oct 12. PMID 29023213
- [Derived] Borghaei H, Paz-Ares L, Horn L, Spigel DR, Steins M, Ready NE, Chow LQ, Vokes EE, Felip E, Holgado E, Barlesi F, Kohlhaufl M, Arrieta O, Burgio MA, Fayette J, Lena H, Poddubskaya E, Gerber DE, Gettinger SN, Rudin CM, Rizvi N, Crino L, Blumenschein GR Jr, Antonia SJ, Dorange C, Harbison CT, Graf Finckenstein F, Brahmer JR. Nivolumab versus Docetaxel in Advanced Nonsquamous Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Oct 22;373(17):1627-39. doi: 10.1056/NEJMoa1507643. Epub 2015 Sep 27. PMID 26412456
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab: Nivolumab 3 mg/kg solution administered intravenously every 2 weeks. Eligible participants transitioned to nivolumab 480 mg every 4 weeks. Participants treated until disease progression, discontinuation due to toxicity, withdrawal of consent or end of study.
- Docetaxel: Docetaxel 75mg/m^2 solution administered intravenously every 3 weeks. Eligible participants transitioned to nivolumab 3 mg/kg every 2 weeks or 480 mg every 4 weeks. Participants treated until disease progression, discontinuation due to toxicity, withdrawal of consent or end of study.
Period: Randomization
Arm/Group | Nivolumab | Docetaxel
Started (Started = Randomized) | 292 | 290
Completed (Completed = Received treatment) | 287 | 268
Not Completed | 5 | 22
Not completed — Adverse event unrelated to study drug | 1 | 0
Not completed — Participant request to discontinue study treatment | 0 | 4
Not completed — Withdrawal by participant | 0 | 12
Not completed — Lost to Follow-up | 0 | 1
Not completed — Participant no longer meets study criteria | 4 | 5
Period: Treatment
Arm/Group | Nivolumab | Docetaxel
Started (Started = Received treatment) | 287 | 268
Participants Who Transitioned to Nivolumab 3 mg/kg | 0 | 17
Participants Who Transitioned to Nivolumab 480 mg | 15 | 1
Completed (Completed = Completed treatment period) | 2 | 0
Not Completed | 285 | 268
Not completed — Disease Progression | 208 | 178
Not completed — Study Drug Toxicity | 23 | 43
Not completed — Death | 2 | 3
Not completed — Adverse event unrelated to study drug | 23 | 10
Not completed — Participant request to discontinue study treatment | 7 | 17
Not completed — Withdrawal by participant | 5 | 5
Not completed — Maximum clinical benefit | 1 | 10
Not completed — Participant no longer meets study criteria | 2 | 0
Not completed — Administrative reason by sponsor | 3 | 0
Not completed — Other reason | 11 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab | Docetaxel | Total
Number analyzed (Participants) | 292 | 290 | 582
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (9.27) | 62.3 (9.75) | 61.6 (9.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 122 | 263
  Male | 151 | 168 | 319
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 9 | 8 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 7 | 9 | 16
  White | 267 | 266 | 533
  Other | 8 | 6 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 16 | 35
  Not Hispanic or Latino | 135 | 141 | 276
  Not Reported | 138 | 133 | 271

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) Time in Months for All Randomized Participants at Primary Endpoint
Description: Overall survival was defined as the time from randomization to the date of death. A participant who has not died will be censored at last known date alive. OS will be followed continuously while participants are on the study drug and every 3 months via in-person or phone contact after participants discontinue the study drug. Median and hazard ratio computed using Kaplan-Meier method.
Time Frame: Randomization until 413 deaths, up to March 2015 (approximately 29 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 292 | 290
Months | 12.19 [9.66 to 14.98] | 9.36 [8.05 to 10.68]
Statistical Analysis 1: Comparison: Nivolumab vs Docetaxel; Test type: Superiority; p = 0.0015, Log Rank; Hazard Ratio (HR) = 0.73, 95.92% CI 2-sided [0.59 to 0.89] — HR = Nivolumab over docetaxel

2. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants whose Best Overall Response (BOR) was a confirmed Complete Response (CR) or Partial Response (PR). BOR was defined as the best investigator-assessed response designation, recorded between the date of randomization and the date of objectively documented progression per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) or the date of subsequent anti-cancer therapy (excluding on-treatment palliative radiotherapy of non-target bone lesions or Central Nervous System (CNS) lesions), whichever occurred first. CR = Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR = At least a 30% decrease in the sum of diameters of target lesions, taking, as reference, the baseline sum diameters. CR+PR, confidence interval based on the Clopper and Pearson method.
Time Frame: From randomization to date of objectively documented progression (up to approximately 110 months)
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 292 | 290
Percentage of participants | 19.5 [15.1 to 24.5] | 12.8 [9.1 to 17.2]

3. Secondary Outcome: Time To Objective Response (TTOR)
Description: Time to Objective Response for participants demonstrating a response (either CR or PR) was defined as the time from the date of randomization to the date of the first confirmed response. CR = Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.; PR = At least a 30% decrease in the sum of diameters of target lesions, taking, as reference, the baseline sum diameters.
Time Frame: From randomization to the date of first confirmed response (up to approximately 110 months)
Population: All randomized participants who demonstrate partial response (PR) or complete response (CR)
Measure: Median (Full Range); unit: Months
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 57 | 37
Months | 2.10 [1.2 to 34.6] | 2.73 [1.4 to 31.2]

4. Secondary Outcome: Duration of Objective Response (DOOR)
Description: DOR was defined as the time from the date of first confirmed response to the date of the first documented tumor progression (per RECIST v1.1), as determined by the investigator, or death due to any cause, whichever occurred first. DOR was evaluated only for confirmed responders (i.e. participants with confirmed CR or PR). CR = Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.; PR = At least a 30% decrease in the sum of diameters of target lesions, taking, as reference, the baseline sum diameters. Participants who neither progressed nor died were censored on the date of their last evaluable tumor assessment. Median computed using Kaplan-Meier method.
Time Frame: From randomization to date of first documented tumor progression or death due to any cause, whichever occurred first (up to approximately 110 months)
Population: All randomized participants who demonstrate partial response (PR) or complete response (CR)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 57 | 37
Months | 17.15 [10.78 to 30.75] | 5.55 [4.40 to 7.03]

5. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from randomization to the date of the first documented tumor progression (per RECIST 1.1) or death due to any cause. Participants who died without a reported prior progression were considered to have progressed on the date of their death. Progression will be assessed every 6 weeks (from the first on-study radiographic assessment) until disease progression is noted. Progressive disease was defined as least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression. Median computed using the Kaplan-Meier method.
Time Frame: From randomization to first confirmed response to the date of the first documented tumor progression or death due to any cause, whichever occurred first (up to approximately 110 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 292 | 290
Months | 2.33 [2.17 to 3.32] | 4.44 [3.45 to 4.86]

6. Secondary Outcome: Percentage of Participants Experiencing Disease-Related Symptom Improvement by Week 12
Description: Disease-related symptom improvement rate by Week 12 was defined as the percentage of randomized participants who had a 10 point or greater decrease from baseline in average symptom burden index score at any time between randomization and Week 12. The participant portion of the Lung Cancer Symptom Scale (LCSS) consisted of 6 symptom-specific questions that addressed cough, dyspnea, fatigue, pain, hemoptysis, and anorexia, plus 3 summary items on symptom distress, interference with activity level, and global health-related Quality of Life (QoL). The scores range from 0 to 100, with 0 representing the best possible score and 100 being the worst possible score. The average symptom burden index score at each assessment was defined as the mean of the 6 symptom-specific questions of the LCSS. 95% CIs were computed using Clopper-Pearson Method.
Time Frame: Randomization to Week 12
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 292 | 290
Percentage of participants | 17.8 [13.6 to 22.7] | 19.7 [15.2 to 24.7]

7. Secondary Outcome: Overall Survival (OS) by PD-L1 Expression at Baseline
Description: Overall survival was defined as the time from randomization to the date of death. A participant who has not died will be censored at last known date alive. Overall Survival time was measured in months for all randomized participants grouped by their baseline PD-L1 expression level. PD-L1 expression in participants was defined as the percent of disease tumor cells demonstrating plasma membrane PD-L1 staining of any intensity using an immunohistochemistry (IHC) assay. Median computed using the Kaplan-Meier method.
Time Frame: From randomization to the date of death or last known date alive (up to approximately 110 months)
Population: All randomized participants who had a tumor biopsy assessed for PD-L1 expression
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 231 | 224
Months
  Participants with baseline PD-L1 expression ≥ 5%: number analyzed (Participants) | 94 | 86
  Participants with baseline PD-L1 expression ≥ 5% | 19.91 [15.08 to 26.12] | 8.11 [6.47 to 10.05]
  Participants with baseline PD-L1 expression < 5%: number analyzed (Participants) | 137 | 138
  Participants with baseline PD-L1 expression < 5% | 9.86 [6.93 to 12.81] | 10.28 [8.54 to 11.96]

8. Secondary Outcome: Objective Response Rate (ORR) by PD-L1 Expression at Baseline
Description: ORR was defined as the percentage of all randomized participants whose Best Overall Response (BOR) was a confirmed Complete Response (CR) or Partial Response (PR). CR = Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.; PR = At least a 30% decrease in the sum of diameters of target lesions, taking, as reference, the baseline sum diameters. CR+PR, confidence interval based on the Clopper and Pearson method. ORR was reported for all randomized participants grouped by their baseline PD-L1 expression level. PD-L1 expression in participants was defined as the percent of disease tumor cells demonstrating plasma membrane PD-L1 staining of any intensity using an immunohistochemistry (IHC) assay.
Time Frame: From randomization to date of objectively documented progression (up to approximately 110 months)
Population: All randomized participants who had a tumor biopsy assessed for PD-L1 expression
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 231 | 224
Percentage of participants
  Participants with baseline PD-L1 expression ≥ 5%: number analyzed (Participants) | 94 | 86
  Participants with baseline PD-L1 expression ≥ 5% | 36.2 [26.5 to 46.7] | 12.8 [6.6 to 21.7]
  Participants with baseline PD-L1 expression < 5%: number analyzed (Participants) | 137 | 138
  Participants with baseline PD-L1 expression < 5% | 10.9 [6.3 to 17.4] | 14.5 [9.1 to 21.5]

9. Post Hoc Outcome: Overall Survival (OS) - Extended Collection
Description: Overall survival was defined as the time from randomization to the date of death. A participant who has not died will be censored at last known date alive. OS will be followed continuously while participants are on the study drug and every 3 months via in-person or phone contact after participants discontinue the study drug. Median computed using Kaplan-Meier method. Note: This outcome measure represents an updated version of the primary endpoint to include additional data collection that has occurred after the primary completion date. (Assessments were made until December 17, 2021).
Time Frame: From randomization to the date of death or last known date alive (up to approximately 110 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 292 | 290
Months | 12.21 [9.66 to 15.08] | 9.49 [8.11 to 10.74]

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from randomization until study completion (up to approximately 110 months). SAEs and Other AEs were assessed from first dose to 100 days after last dose of study therapy (up to approximately 108 months).
Description: All-Cause Mortality = all randomized participants. Serious Adverse Events and Other Adverse Events = all treated participants.
  ARM 1: AEs that occurred on 3 mg/kg Nivolumab, ARM 2: AEs that occurred on 480 mg Nivolumab, ARM 3: AEs that occurred on Docetaxel treatment only, ARM 4: Extension phase of Docetaxel arm: AEs that occurred on 3 mg/kg Nivolumab, ARM 5: Extension phase of Docetaxel arm: AEs that occurred on or 480 mg Nivolumab.
Groups:
- Nivolumab 3 mg/kg: Nivolumab 3 mg/kg solution administered intravenously every 2 weeks. Participants treated until disease progression, discontinuation due to toxicity, withdrawal of consent or end of study.
- Nivolumab 480 mg: Nivolumab 480 mg solution administered intravenously every 4 weeks. Participants treated until disease progression, discontinuation due to toxicity, withdrawal of consent or end of study.
- Docetaxel: Docetaxel 75mg/m^2 solution administered intravenously every 3 weeks. Participants treated until disease progression, discontinuation due to toxicity, withdrawal of consent or end of study.
- Extension Phase of Docetaxel Arm: Nivolumab 3 mg/kg: Eligible participants from the Docetaxel arm who transitioned to nivolumab 3 mg/kg every 2 weeks via extension phase. Participants treated until disease progression, discontinuation due to toxicity, withdrawal of consent or end of study.
- Extension Phase of Docetaxel Arm: Nivolumab 480 mg: Eligible participants from the Docetaxel arm who transitioned to nivolumab 480 mg every 4 weeks via extension phase. Participants treated until disease progression, discontinuation due to toxicity, withdrawal of consent or end of study.
Arm/Group | Nivolumab 3 mg/kg | Nivolumab 480 mg | Docetaxel | Extension Phase of Docetaxel Arm: Nivolumab 3 mg/kg | Extension Phase of Docetaxel Arm: Nivolumab 480 mg
All-Cause Mortality (participants affected / at risk) | 258/292 | 2/15 | 266/290 | 14/17 | 0/1
Serious Adverse Events (participants affected / at risk) | 172/287 | 5/15 | 161/268 | 9/17 | 1/1
Other Adverse Events (participants affected / at risk) | 267/287 | 12/15 | 258/268 | 12/17 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab 3 mg/kg (N=287) | Nivolumab 480 mg (N=15) | Docetaxel (N=268) | Extension Phase of Docetaxel Arm: Nivolumab 3 mg/kg (N=17) | Extension Phase of Docetaxel Arm: Nivolumab 480 mg (N=1)
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 4 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 24 | 0 | 0
Haematotoxicity (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 8 | 0 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 2 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 2 | 0 | 3 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Retinal tear (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 3 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 0 | 4 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0
Asthenia (General disorders) | 3 | 0 | 3 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
Complication associated with device (General disorders) | 1 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 3 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 2 | 1 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 2 | 0 | 4 | 1 | 0
Inflammation (General disorders) | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 3 | 0 | 1 | 0 | 0
Pain (General disorders) | 4 | 0 | 4 | 0 | 0
Pyrexia (General disorders) | 6 | 0 | 4 | 0 | 0
Sudden death (General disorders) | 2 | 0 | 3 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 5 | 1 | 5 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 2 | 1 | 0 | 0 | 0
Encephalitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Febrile infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Fungal oesophagitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 2 | 0 | 2 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lung abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Nail infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 22 | 1 | 18 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Pneumonia mycoplasmal (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia necrotising (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Post procedural pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0 | 3 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Spontaneous bacterial peritonitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Vascular device infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0
General physical condition abnormal (Investigations) | 2 | 0 | 2 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 6 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 4 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 58 | 0 | 40 | 2 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 3 | 0 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0 | 10 | 0 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Central nervous system necrosis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 4 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Hemiplegia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
IVth nerve paresis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 2 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 3 | 0 | 0
Panic attack (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 1 | 8 | 0 | 0
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10 | 0 | 4 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 13 | 0 | 5 | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 | 0 | 4 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 2 | 0 | 0
Embolism (Vascular disorders) | 1 | 0 | 2 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Peripheral artery occlusion (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Peripheral artery stenosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab 3 mg/kg (N=287) | Nivolumab 480 mg (N=15) | Docetaxel (N=268) | Extension Phase of Docetaxel Arm: Nivolumab 3 mg/kg (N=17) | Extension Phase of Docetaxel Arm: Nivolumab 480 mg (N=1)
Anaemia (Blood and lymphatic system disorders) | 37 | 0 | 68 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 29 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 82 | 0 | 0
Hypothyroidism (Endocrine disorders) | 21 | 0 | 0 | 2 | 0
Lacrimation increased (Eye disorders) | 3 | 0 | 22 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 19 | 0 | 16 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 11 | 0 | 14 | 1 | 0
Constipation (Gastrointestinal disorders) | 69 | 2 | 50 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 57 | 2 | 74 | 2 | 0
Nausea (Gastrointestinal disorders) | 72 | 2 | 85 | 4 | 0
Stomatitis (Gastrointestinal disorders) | 8 | 0 | 24 | 1 | 0
Vomiting (Gastrointestinal disorders) | 44 | 3 | 30 | 1 | 0
Asthenia (General disorders) | 60 | 1 | 63 | 1 | 0
Fatigue (General disorders) | 96 | 0 | 104 | 7 | 0
Mucosal inflammation (General disorders) | 6 | 0 | 19 | 1 | 0
Non-cardiac chest pain (General disorders) | 17 | 0 | 18 | 0 | 0
Oedema peripheral (General disorders) | 36 | 0 | 46 | 1 | 0
Pain (General disorders) | 21 | 0 | 19 | 0 | 0
Pyrexia (General disorders) | 37 | 0 | 44 | 1 | 0
Nasopharyngitis (Infections and infestations) | 14 | 2 | 11 | 1 | 0
Pneumonia (Infections and infestations) | 9 | 2 | 16 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 19 | 1 | 13 | 2 | 0
Alanine aminotransferase increased (Investigations) | 20 | 1 | 6 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 14 | 1 | 3 | 0 | 0
Neutrophil count decreased (Investigations) | 2 | 0 | 18 | 0 | 0
Weight decreased (Investigations) | 28 | 0 | 21 | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 22 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 91 | 0 | 64 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 15 | 0 | 15 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 72 | 3 | 41 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 45 | 2 | 18 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 18 | 0 | 14 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 15 | 0 | 8 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 20 | 2 | 35 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 29 | 1 | 30 | 1 | 0
Dizziness (Nervous system disorders) | 30 | 1 | 25 | 1 | 0
Dysgeusia (Nervous system disorders) | 6 | 0 | 20 | 0 | 1
Headache (Nervous system disorders) | 33 | 1 | 35 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 12 | 0 | 28 | 2 | 0
Paraesthesia (Nervous system disorders) | 14 | 0 | 25 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 7 | 0 | 14 | 1 | 0
Anxiety (Psychiatric disorders) | 18 | 0 | 8 | 0 | 0
Insomnia (Psychiatric disorders) | 25 | 2 | 23 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 83 | 5 | 67 | 6 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 68 | 1 | 64 | 6 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 11 | 0 | 19 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 16 | 0 | 15 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 14 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 | 1 | 16 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 16 | 1 | 10 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 11 | 0 | 70 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 24 | 0 | 9 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 7 | 1 | 18 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 37 | 1 | 7 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 41 | 3 | 18 | 2 | 0
Hypertension (Vascular disorders) | 14 | 2 | 4 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 3 | 0 | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 0 | 3 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 3 | 0 | 1 | 1 | 0
Tachycardia (Cardiac disorders) | 6 | 0 | 8 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 1 | 1 | 0 | 0
Excessive cerumen production (Ear and labyrinth disorders) | 2 | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 2 | 0 | 3 | 1 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 4 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 7 | 0 | 12 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 7 | 1 | 8 | 1 | 0
Chest discomfort (General disorders) | 2 | 1 | 1 | 0 | 0
Chest pain (General disorders) | 11 | 1 | 6 | 1 | 0
Influenza like illness (General disorders) | 3 | 0 | 3 | 1 | 1
Nodule (General disorders) | 1 | 1 | 1 | 0 | 0
Swelling (General disorders) | 1 | 1 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 10 | 2 | 7 | 0 | 0
Campylobacter infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Candida infection (Infections and infestations) | 1 | 0 | 5 | 1 | 0
Conjunctivitis (Infections and infestations) | 6 | 1 | 4 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 3 | 0 | 3 | 1 | 0
Respiratory tract infection (Infections and infestations) | 5 | 0 | 3 | 1 | 0
Sinusitis (Infections and infestations) | 13 | 1 | 3 | 0 | 0
Urinary tract infection (Infections and infestations) | 13 | 0 | 9 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 5 | 1 | 1 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 1 | 1 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 7 | 1 | 6 | 0 | 0
Blood creatinine increased (Investigations) | 11 | 0 | 4 | 1 | 0
Blood glucose increased (Investigations) | 2 | 1 | 6 | 0 | 0
Blood magnesium decreased (Investigations) | 1 | 0 | 1 | 1 | 0
Haemoglobin decreased (Investigations) | 5 | 1 | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Weight increased (Investigations) | 11 | 0 | 5 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 6 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 9 | 1 | 7 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 10 | 1 | 4 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 1 | 3 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 11 | 1 | 6 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 8 | 1 | 4 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 12 | 1 | 4 | 0 | 0
Memory impairment (Nervous system disorders) | 2 | 1 | 1 | 0 | 0
Motor dysfunction (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 10 | 1 | 5 | 0 | 0
Depression (Psychiatric disorders) | 8 | 0 | 10 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 2 | 1 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 2 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 4 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 2 | 1 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 9 | 1 | 5 | 0 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Haematoma (Vascular disorders) | 1 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 7 | 1 | 1 | 0 | 0
Hypotension (Vascular disorders) | 12 | 1 | 9 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.